CLINICAL TRIAL: NCT04624074
Title: Pilot Testing a TMCU Adapted for Young Adults With First Episode Psychosis
Brief Title: Pilot Testing the Check Up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Melanie E Bennett, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01MH120550-01A1 (NIH)
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Cannabis Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teen Marijuana Checkup - adapted (Experimental): Teen Marijuana Checkup will be adapted for youth and young adults with first episode psychosis. The Teen Marijuana Checkup includes two intervention sessions. In Session 1, the interventionist uses motivational interviewing skills to hear the adolescent's history and current concerns with marijuana. The personalized feedback report generated from the baseline assessment is reviewed. In Session 2, the interventionist elicits change talk and guides discussion on making changes to reduce or stop marijuana use.
  Interventions: Behavioral: Teen Marijuana Check Up

INTERVENTIONS:
Behavioral: Teen Marijuana Check Up — Teen Marijuana Checkup will be adapted for youth and young adults with first episode psychosis. The Teen Marijuana Checkup includes two intervention sessions. In Session 1, the interventionist uses motivational interviewing skills to hear the adolescent's history and current concerns with marijuana. The personalized feedback report generated from the baseline assessment is reviewed. In Session 2, the interventionist elicits change talk and guides discussion on making changes to reduce or stop marijuana use.

SUMMARY:
We propose to pilot test an adapted version of the Teen Marijuana Check Up (TMCU) for persistent cannabis users with first episode psychosis (FEP) in Coordinated Specialty Care (CSC). The adapted version of the TMCU will include tailoring to risks of persistent cannabis use in FEP, providing education on lower risk cannabis use, and adding a session to address collaborative planning to maintain CSC engagement and antipsychotic adherence and to reduce harm associated with cannabis use.

DETAILED DESCRIPTION:
We propose to adapt the Teen Marijuana Check Up for persistent cannabis users with FEP in CSC. Dr. Walker, the developer of the TMCU, will be a consultant. Adaptations will include tailoring content of assessment and feedback to risks of persistent cannabis use in FEP, providing education on lower risk cannabis use, and adding a session to address collaborative planning to maintain CSC engagement and antipsychotic adherence and to reduce harm associated with cannabis use. We will also develop guidelines for integrating continued collaborative, harm-reduction focused discussion of cannabis use into CSC, consider adding booster or check-in sessions, and specify how family members can be brought into the check-up process. To inform these adaptations, we will collect quantitative data from cannabis-using FEP patients (n of 40) and conduct qualitative interviews with cannabis-using patients, family members, and CSC clinicians (15 of each) about their perspectives on cannabis use and CSC participation (Aim 1). We will use these data as part of an iterative process to specify the adapted intervention that will integrate information gathered from team discussion and focus groups with FEP patients and family members and vetting of intervention components by key stakeholders (Aim 2). Finally, we will conduct a pilot of the adapted intervention (n of 40 cannabis-using FEP patients compared to matched controls) to examine feasibility, acceptability, fidelity, and preliminary impact on intervention targets and outcomes (Aim 3). If results are promising, the intervention can be tested in a large RCT across the EPINET.

ELIGIBILITY:
Inclusion Criteria:

1. Age 13-35
2. DSM-5 diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, brief psychotic disorder, delusional disorder, other specified schizophrenia spectrum and other psychotic disorder, and unspecified schizophrenia spectrum and other psychotic disorder
3. Duration of illness: ≤ 2 years
4. Enrolled at a Coordinated Specialty Care program
5. Report current use of cannabis
6. Ability and willingness to provide informed consent to participate

Exclusion Criteria:

1. Individuals who do not meet all inclusion criteria are excluded.

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Timeline Followback | baseline, immediately after the intervention
  Change in cannabis use
Modified Colorado Symptom Index | baseline, immediately after the intervention
  Change in psychosis symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No